CLINICAL TRIAL: NCT06995378
Title: Patient-Centered Lab Result Communication Tool for Older Adults With Elevated Hemoglobin A1c (A1c) or Chronic Kidney Disease (CKD)
Brief Title: Patient-centered Precision Medicine Lab Result Communication for Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P30AG073104 (NIH); P30AG073104 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-05

CONDITIONS: Kidney Disease, Chronic
Keywords: lab result; lab result communication tool
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Lab Result Arm (Experimental): Participants (patients aged 65+ and UCLA Health providers) will engage in a tool integrated into the EHR system to personalize how lab results are communicated to patients aged 65+ and their providers. The tool uses individual risk information and different visual/text formats to display results. Participants will view the tool and access user experience through observation, interviews, and surveys.
  Interventions: Behavioral: Lab Result Communication Tool

INTERVENTIONS:
Behavioral: Lab Result Communication Tool — A behavioral intervention delivered through a personalized EHR-integrated lab result communication tool designed to improve emotional and cognitive responses to lab results among adults aged 65+. The tool applies behavioral science principles such as risk personalization, simplified messaging, and visual framing to reduce patient anxiety, enhance understanding, and support informed decision-making.

SUMMARY:
For adults >65 years and their providers, the investigators will test the usability and design of a tool to replace standard uniform reporting of lab results to patients and their providers with a new personalized EHR lab result communication tool that: 1) extracts patient-level data from the EHR; 2) calculates individual risk; and 3) for patients with very low risk, communicates the individualized risk information. The investigators will employ a range of user experience research methods to understand how patient and provider users interact with the new lab result communication tool and to assess their comprehension of the lab results.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria: Older adults (aged >65 years) with a UCLA primary care provider who are:

* Enrolled in the patient portal;
* English-speaking (as the language of the tool is currently only in English, and it would be impractical to have validated translations created for all of the potential variations and derivatives of the tool mock-ups); and
* Without dementia or other neurocognitive disease.

Provider Inclusion Criteria:

-UCLA Health providers who care for large numbers of older adults in outpatient settings.

Exclusion Criteria:

Patient Exclusion Criteria:

* Have lab results outside of the defined inclusion ranges;
* Do not have a UCLA PCP;
* Are under the age of 65;
* Are not English speaking (as the tool prototypes are only in English until final verbiage is determined);
* Are not enrolled in the UCLA MyChart patient portal; or
* Are diagnosed with dementia

Provider Exclusion Criteria:

-Do not care for large numbers of older adults in outpatient settings

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported anxiety about lab results after using the personalized tool | Immediately after the user experience session
  Participants will complete a structured post-session survey using a 5-point Likert scale titled "Emotional Response to Lab Results". The scale ranges from 1 (Strongly Disagree) to 5 (Strongly Agree). Higher scores indicate lower anxiety and greater emotional reassurance. Survey items will assess their emotional response, including levels of anxiety and reassurance, after viewing lab results through the new tool. Responses will be compared to participants' recalled or expected emotional responses based on past experiences with standard lab result communication formats.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No